CLINICAL TRIAL: NCT06067555
Title: Characterization of Immune Response to Intradermal Influenza Vaccination
Brief Title: Intradermal Influenza Vaccination
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Chan Zuckerberg Initiative (Other); National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH); Silicon Valley Community Foundation (Other); University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2000035891; 2T32AR007016-47 (NIH)
Record Dates: First submitted 2023-09-27; First posted 2023-10-05 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Vaccine Reaction

STUDY DESIGN:
Intervention Model Description: In the first year, a total of 39 participants will be enrolled (5 for most cohorts; 3 for each saline control group).
  After preliminary analysis of the first season, we will choose the two most informative skin biopsy time points (2 hour, 6 hour, Day 1, Day 3, or Day 28) and plan for expansion of these cohorts in subsequent influenza seasons for a total of 100 participants per intradermal influenza vaccination cohort. An IM-control group of N=5 will be kept for each flu season; Therefore the total number of participants will be 249 participants. We will not include saline controls in subsequent seasons.
  Participants in saline-control cohorts will be restricted from obtaining flu vaccination until after Day 28; after Day 28, they will be allowed to receive influenza vaccination at their discretion. We will ask and record if and when they received vaccination.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (9):
- Intramuscular (IM) Control (Active Comparator): An intramuscular control group, from which no skin biopsies will be taken after vaccination. Only the intramuscular cohort will receive the flu vaccine via standard IM route in the deltoid region of the upper arm.
  Interventions: Biological: Fluzone® Quadrivalent
- ID-2hour (Experimental): Participants receive intradermal flu vaccination in the upper arm and will have skin biopsy of vaccination site 2 hours after vaccine administration.
  Interventions: Device: MicronJet; Biological: Fluzone® Quadrivalent
- ID-6hour (Experimental): Participants receive intradermal flu vaccination in the upper arm and will have skin biopsy of vaccination site 6 hours after vaccine administration.
  Interventions: Device: MicronJet; Biological: Fluzone® Quadrivalent
- ID-1day (Experimental): Participants receive intradermal flu vaccination in the upper arm and will have skin biopsy of vaccination site 1 day after vaccine administration.
  Interventions: Device: MicronJet; Biological: Fluzone® Quadrivalent
- ID-3day (Experimental): Participants receive intradermal flu vaccination in the upper arm and will have skin biopsy of vaccination site 3 days after vaccine administration.
  Interventions: Device: MicronJet; Biological: Fluzone® Quadrivalent
- ID-28day (Experimental): Participants receive intradermal flu vaccination in the upper arm and will have skin biopsy of vaccination site 3 days after vaccine administration.
  Interventions: Device: MicronJet; Biological: Fluzone® Quadrivalent
- Sal-2hour (Placebo Comparator): A control group in which bacteriostatic saline is injected intradermally in lieu of influenza vaccine. A skin biopsy will be taken from the "vaccination" site 2 hours after administration.
  Interventions: Device: MicronJet; Other: Bacteriostatic Saline
- Sal-6hour (Placebo Comparator): A control group in which bacteriostatic saline is injected intradermally in lieu of influenza vaccine. A skin biopsy will be taken from the "vaccination" site 6 hours after administration.
  Interventions: Device: MicronJet; Other: Bacteriostatic Saline
- Sal-1hour (Placebo Comparator): A control group in which bacteriostatic saline is injected intradermally in lieu of influenza vaccine. A skin biopsy will be taken from the "vaccination" site 1 day after administration.
  Interventions: Device: MicronJet; Other: Bacteriostatic Saline

INTERVENTIONS:
Device: MicronJet — MicronJet 600 syringe will be used to administer intradermal flu vaccine injections
  Arms: ID-1day; ID-28day; ID-2hour; ID-3day; ID-6hour; Sal-1hour; Sal-2hour; Sal-6hour
Biological: Fluzone® Quadrivalent — Intradermal injections of 0.3mL
  Arms: ID-1day; ID-28day; ID-2hour; ID-3day; ID-6hour
Biological: Fluzone® Quadrivalent — Intramuscular injection of 0.3mL
  Arms: Intramuscular (IM) Control
Other: Bacteriostatic Saline — Intradermal injection of 0.3mL (control)
  Arms: Sal-1hour; Sal-2hour; Sal-6hour

SUMMARY:
The goal of this study is to characterize the immune response, both innate and adaptive, as well as locally and systemic, to intradermal (ID) vaccination in healthy individuals. The intervention involves intradermal administration of an FDA-approved intramuscular seasonal influenza vaccine, using an FDA-approved device MicronJet. Investigators will measure antibody titers, cell subtypes, and multi-omic profiles, by collecting skin and peripheral blood at baseline and at several time points after vaccination. The primary objective is to identify baseline correlates of immune response in the skin and peripheral blood to the seasonal influenza vaccine. The investigators secondary goals are to describe the inflammatory response in the skin over time.

DETAILED DESCRIPTION:
Subjects will remain on study and may optionally repeat study visits (including vaccination) annually through the 2025-26 influenza season, with final study follow-up up to 1 year after vaccination. Sampling individual subjects across several influenza seasons will allow for monitoring of multi-season responses.

Skin, blood, nasal mucosal lining fluid, nasopharyngeal cells, saliva, and skin microbe samples will be collected at various timepoints before and up to 365 days after vaccination to explore short and long-term effects of immunization. Subjects may optionally provide stool samples.

ELIGIBILITY:
In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study, as well as have deidentified samples and data stored for future research.
3. Able to proficiently speak, read, and write English.
4. Male or female, aged 18-40 years old at time of initial enrollment

   a. Participant is allowed to participate in subsequent influenza seasons even if they will be >40 years old.
5. In good general health as evidenced by medical history

Individuals meeting any of the following criteria will be excluded from study participation:

1. CBC with differential, lymphocyte phenotyping with T, B, and natural killer cells (TBNK), complete metabolic panel, anti-CMV immunoglobulin (Ig) G and IgM, and/or anti-Epstein-Barr virus (EBV) antibody panel values outside of the Yale Department of Laboratory Medicine normal reference ranges and deemed clinically significant by the PI at the time of screening.
2. Positive result for anti-HIV 1/2 antibody screening at the time of screening.
3. Prior receipt of a current seasonal influenza vaccine (for the season of participation).
4. History of allergy or hypersensitivity to any components of the study vaccine (e.g., egg protein).
5. History of severe reactions to vaccines.
6. Use of an oral glucocorticoid within the past 30 days.
7. Receipt of a live-attenuated vaccine within the past 3 months.
8. Receipt of any experimental vaccine.
9. Receipt of any other type of vaccine (non-live and non-experimental, e.g., tetanus, diphtheria, and pertussis [TDaP]) within the past 3 months.
10. Planned vaccination before day 100 after study vaccination.
11. Current or recent use (within the past 90 days) of immunoglobulin therapy.
12. Surgery within the past 8 weeks, or planned surgery before day 28.
13. Current (within the past 30 days) treatment for active malignancy.
14. Cancer chemotherapy in the past 2 years.
15. Administration of any blood products within 90 days of the screening, or planned administration before day 100.
16. History of parasitic, amebic, fungal, or mycobacterial infections within the past 1 year, with the exception of tinea pedis and onychomycosis.
17. History of autoimmune or autoinflammatory disease.

    a. In particular skin-related (i.e. psoriasis, lichen planus, lupus, neutrophilic dermatoses, atopic dermatitis)
18. History of keloids
19. History of a bleeding disorder.
20. Current use (within the past 30 days) of illicit drugs (per subject report), with the exception of marijuana.
21. Current alcohol use disorders (criteria per Diagnostic and Statistical Manual of Mental Disorders, fifth edition), within the past 30 days.
22. Serious, ongoing, uncontrolled infection within the past 30 days as per the judgement of the PI.
23. History of Guillain-Barre syndrome (GBS).
24. BMI ≥ 30.
25. Known or suspected immunodeficiency within 1 year, including documented HIV infection.
26. Pregnancy or planning to become pregnant during the study period. (Women of childbearing potential must have a negative urine or serum pregnancy test at screening.)
27. Presence of conditions that, in the judgment of the PI, may put the individual at undue risk or compromise the scientific objectives of the study.

Co-enrollment guidelines: Co-enrollment in other trials is restricted, other than enrollment on observational studies. Consideration for co-enrollment in trials evaluating the use of a licensed medication will require the approval of the PI. Study staff should be notified of co-enrollment on any other protocol as it may require the approval of the PI.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 249 (Estimated)
Dates: Start 2024-01-24 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Change in antibody titer concentration to vaccination-Blood | Day 0 and Day 28
  Change in antibody titer to vaccination as measured by microneutralization titers at day 0 and day 28 will be correlated with biomarkers in the blood using generalized estimating equations.
Change in antibody titer concentration to vaccination-Skin | Day 0 and Day 28
  Change in antibody titer to vaccination as measured by microneutralization titers at day 0 and day 28 will be correlated with biomarkers in the skin at baseline using generalized estimating equations.

SECONDARY OUTCOMES:
Change in antibody titer concentration to vaccination | Day 0 and Day 28
  Change in antibody titer response to vaccination as measured by microneutralization titers at day 0 and day 28 and its relationship with established baseline biomarkers (CD38+, CD20+, B cell, among others) and post-vaccination biomarkers (plasmablast, among others) in the blood will be correlated using generalized estimating equations.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Johnston, Principal Investigator — Yale University
Locations (1):
- Church Street Research Unit, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
Human data generated in this study will be shared for future research as follows:
  * De-identified data in an NIH-funded or approved public repository, including
    * genetic data in the database of Genotypes and Phenotypes (dbGaP).
    * gene expression and chromatin profiling data in the National Center for Biotechnology Information (NCBI) Gene Expression Omnibus (GEO).
    * sequencing data in the NCBI Sequence Read Archive (SRA).
    * flow cytometry data in FlowRepository.
  * De-identified or identified data with approved outside collaborators under appropriate agreements.
Time Frame: Data will be shared before publication through presentations at meetings and seminars; raw and complete data sets will not be shared until the time of publication or shortly thereafter.